CLINICAL TRIAL: NCT01025349
Title: Retrospective Analysis of Salvage Therapy With Bevacizumab Plus Docetaxel and Cisplatin for Taiwanese Metastatic Breast Cancer
Brief Title: Salvage Therapy With Bevacizumab Plus Docetaxel and Cisplatin for Taiwanese Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Cheng-Jeng Tai, M.D., Director., Section of Hematology-Oncology, Department of Medicine, Taipei Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMUH-01-09-09
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-12

CONDITIONS: Metastatic Breast Cancer
Keywords: bevacizumab; metastatic breast cancer; docetaxel
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- metastatic breast cancer (Experimental): Patients with histological or cytological proven metastatic breast cancer were recruited. The previous hormonal therapy for metastatic breast cancer or cytotoxic therapy was allowed. The Her2/Neu over-expressive status should be negative. Patients with brain metastasis are excluded.
  Interventions: Drug: Bevacizumab, docetaxel, cisplatin

INTERVENTIONS:
Drug: Bevacizumab, docetaxel, cisplatin — Bevacizumab 8 mg/kg(over 60 minutes) on first day of first cycle, followed by 5 mg/kg on first day of the rest cycles, repeat every 2 weeks.
  docetaxel 45 mg/m2(over 60 minutes) on day 1 of each cycle, repeat every 2 weeks.
  cisplatin 50 mg/m2(over 4 hours) on day 1 of each cycle, repeat every 2 weeks.
  Other Names: bevacizumab: avastin; docetaxel: taxotere

SUMMARY:
Bevacizumab is a monoclonal antibody currently used for the treatment of colorectal cancer. It works by preventing the formation of new blood vessels (angiogenesis). The drug has been shown to inhibit vascular endothelial growth factor (VEGF) activity. Previous research showed positive findings in other solid tumors that had metastasized. In this study, the investigators are investigating the response of adding bevacizumab to conventional chemotherapy for metastatic breast cancer patients.

DETAILED DESCRIPTION:
Targeted chemotherapy has gradually become the mainstay of cancer treatment in present day. Targeted medications such as trastuzumab, bevacizumab and lapatinib have recently been more extensively adopted for many cancers, particularly breast cancer. Among these targeted medications, bevacizumab is a monoclonal antibody acting on vascular endothelial growth factor receptor and it works by preventing the formation of new blood vessels (angiogenesis). Published articles indicated that monotherapy of bevacizumab on breast cancer showed only a 9-17% response rate, while combining with paclitaxel, the treatment outcome appeared to improve progression-free survival and the objective response rate. We are curious about the additive effect of bevacizumab on conventional chemotherapy, the toxicities induced when combined target therapy with conventional chemotherapy and the duration of remission that these treatment could achieve. In this study, we utilized bevacizumab, docetaxel plus cisplatin for metastatic breast cancer patients and furthermore, we are evaluated the treatment response, toxicities and duration of remission as our main goals.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2.
* Normal left ventricular ejection fraction (LVEF).
* Age ≤ 65 years.
* At least one unidimensionally measurable lesion by imaging studies.
* AST/ALT 2.5 ULN (< 5 ULN if liver metastases).
* Serum bilirubin 3 ULN, Serum Creatinine 1.5 ULN.
* Urine dipstick of proteinuria <2+.
* Women of childbearing potential must have a negative serum pregnancy test.

Exclusion Criteria:

* Uncontrolled hypertension (systolic blood pressure > 160 mm Hg, diastolic blood pressure > 90 mm Hg).
* Prior exposure to bevacizumab.
* Planned radiotherapy for underlying disease (prior completed radiotherapy treatment allowed), except bone metastasis.
* Evidence of bleeding diathesis or coagulopathy.
* Clinically significant (i.e. active) cardiovascular disease for example cerebrovascular accidents (≤ 6 months), myocardial infarction (≤ 6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication. Stroke in the preceding six months.
* Evidence of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of bevacizumab with chemotherapy.
* Ongoing treatment with aspirin (> 325 mg/day) or other medications known to predispose to gastrointestinal ulceration.
* Pregnancy (positive serum pregnancy test) and lactation. Any other serious or uncontrolled illness which, in the opinion of the investigator, makes it undesirable for the patient to enter the trial.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Response Rate | every 3 months

SECONDARY OUTCOMES:
Time to Progression(TTP), Progression free survival, overall survival, safety, Quality of Life | every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Jeng Tai, M.D., Principal Investigator — Section of Hematology-Oncology, Department of Medicine, Taipei Medical University Hospital
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Miller KD, Sweeney CJ, Sledge GW Jr. Redefining the target: chemotherapeutics as antiangiogenics. J Clin Oncol. 2001 Feb 15;19(4):1195-206. doi: 10.1200/JCO.2001.19.4.1195. PMID 11181686
- [Background] Moy B, Goss PE. Lapatinib: current status and future directions in breast cancer. Oncologist. 2006 Nov-Dec;11(10):1047-57. doi: 10.1634/theoncologist.11-10-1047. PMID 17110623
- [Background] Chu E. Bevacizumab targeted therapy: validation of angiogenesis as a key target for advanced colorectal cancer. Clin Colorectal Cancer. 2004 May;4(1):16. doi: 10.3816/ccc.2004.n.006. No abstract available. PMID 15207014
- [Background] Eniu A. Integrating biological agents into systemic therapy of breast cancer: trastuzumab, lapatinib, bevacizumab. J BUON. 2007 Sep;12 Suppl 1:S119-26. PMID 17935269
- [Background] Caprioni F, Fornarini G. Bevacizumab in the treatment of metastatic colorectal cancer. Future Oncol. 2007 Apr;3(2):141-8. doi: 10.2217/14796694.3.2.141. PMID 17381413
- [Background] Jubb AM, Hurwitz HI, Bai W, Holmgren EB, Tobin P, Guerrero AS, Kabbinavar F, Holden SN, Novotny WF, Frantz GD, Hillan KJ, Koeppen H. Impact of vascular endothelial growth factor-A expression, thrombospondin-2 expression, and microvessel density on the treatment effect of bevacizumab in metastatic colorectal cancer. J Clin Oncol. 2006 Jan 10;24(2):217-27. doi: 10.1200/JCO.2005.01.5388. Epub 2005 Dec 19. PMID 16365183
- [Background] Link JS, Waisman JR, Nguyen B, Jacobs CI. Bevacizumab and albumin-bound paclitaxel treatment in metastatic breast cancer. Clin Breast Cancer. 2007 Oct;7(10):779-83. doi: 10.3816/CBC.2007.n.039. PMID 18021479